CLINICAL TRIAL: NCT00927446
Title: Endoscopy Screening for Esophageal Neoplasm With Narrow Band Imaging in Patients With Head and Neck Cancer: A Controlled Tandem Endoscopy Trial
Brief Title: Endoscopy Screening for Esophageal Cancer
Status: Terminated | Type: Observational
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Hsing-Hong Chen/Superintendent, Lotung Poh-Ai hospital
Other Study IDs: OMCP-98-006
Record Dates: First submitted 2009-06-22; First posted 2009-06-25 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Head and Neck Cancer
Keywords: esophageal cancer; head and neck cancer; narrow band imaging; endoscopy; screening
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — endoscopic biopsy for histopathological examination
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endoscopy screening: Patients with tissue diagnosis of head and neck cancer undergo endoscopy screening with conventional white light system first. Then the entire esophagus is examined under the NBI system by another endoscopist, who is blinded to the result of the conventional endoscopy.
  Interventions: Procedure: Endoscopy screening with narrow band imaging

INTERVENTIONS:
Procedure: Endoscopy screening with narrow band imaging — Narrow Band Imaging (NBI) system, an optical technology that enhances the visualization of superficial vascular network, may be superior to the conventional white light endoscopy for the detection of neoplastic lesions.
  Other Names: NBI

SUMMARY:
Patients with head and neck cancer frequently develop synchronous or metachronous esophageal malignancies. Previous studies have demonstrated the efficacy of endoscopic screening for esophageal cancer in head and neck cancer patients. The Narrow Band Imaging (NBI) system, an optical technology that enhances the visualization of superficial vascular network, may be superior to the conventional white light endoscopy for the detection of neoplastic lesions. However, whether the application of NBI improves the detection results have not been critically evaluated.

This study aims to investigate the diagnostic value of the NBI system in the endoscopic screening for esophageal neoplastic lesions in patients with head and neck cancer.

DETAILED DESCRIPTION:
This is a prospective blinded controlled tandem endoscopy trial conducted in a regional medical center (Lotung Poh-Ai Hospital, Taiwan). Patients with tissue diagnosis of head and neck cancer are enrolled. Endoscopy screening for esophageal lesions is first performed by using the conventional white light system. Suspicious lesions are recorded. Then the entire esophagus is examined under the NBI system by another endoscopist, who is blinded to the result of the conventional endoscopy. After the endoscopic inspection completed, all suspicious lesions are biopsied. Before each procedure, which one of the two participating endoscopists applies the conventional or NBI system is randomized. The diagnostic rate of esophageal neoplasm by the conventional white light system and that of the NBI system are compared.

The endpoint is the neoplastic lesion detected on endoscopic biopsy. We considered invasive cancer, carcinoma in-situ, and high-grade dysplasia (which usually cannot be distinguished from carcinoma in situ) as the primary points. Any dysplastic lesions were considered as secondary points.

ELIGIBILITY:
Inclusion Criteria:

* patients with tissue diagnosis of head and neck cancer
* histopathology of head and neck cancer is carcinoma (including squamous cell carcinoma, adenocarcinoma or undifferentiated)
* aged more than 18 years old
* agree to under go upper gastrointestinal endoscopy

Exclusion Criteria:

* lack of written informed consent
* the origin of head and neck cancer is metastatic
* histopathology of head and neck cancer is not carcinoma (e.g., sarcoma, lymphoma, etc)
* incomplete upper gastrointestinal endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tissue diagnosis of head and neck carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pathological interpretation of biopsy specimen for invasive cancer, carcinoma in-situ, or high-grade dysplasia | Within 3 days of endoscopy examination

SECONDARY OUTCOMES:
Pathological interpretation of biopsy specimen for any grade of dysplasia | within 3 days of endoscopy examination

CONTACTS AND LOCATIONS:
Overall Officials: Tzeng-Huey Yang, M.D., Principal Investigator — Lotung Poh-Ai Hospital
Locations (1):
- Lotung Poh-Ai Hospital, Yilan, Taiwan